CLINICAL TRIAL: NCT06917495
Title: Rifapentine- And Moxifloxacin-Containing Short-Course Regimens for Mild Spinal Tuberculosis: A Multicenter, Randomized, Non-inferiority Clinical Trial
Brief Title: Short-Course Anti-tuberculosis Regimens for Mild Spinal Tuberculosis
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shandong University (Other)
Collaborators: Shandong Public Health Clinical Center (Other Government)
Responsible Party: Principal Investigator, Wei Zhao, Head of department of clinical pharmacy and pharmacology, Shandong University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SDU-2024-RPT-003
Record Dates: First submitted 2025-03-25; First posted 2025-04-08 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-03

CONDITIONS: Mild Spinal Tuberculosis
MeSH Terms: interventions — Rifampin; Isoniazid; rifapentine; Moxifloxacin; Pyrazinamide; Ethambutol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Empirical long course regimen (Active Comparator): Drug: Rifampicin, once daily, 600 mg, administered for 52 weeks. Drug: Isoniazid, once daily, 300 mg, administered for 52 weeks. Drug: Pyrazinamide, once daily, dosage adjusted based on body weight: 1000 mg for < 55 kg, 1500 mg for ≥ 55-75 kg, and 2000 mg for > 75 kg, administered for the first 8 weeks.
  Drug: Ethambutol, once daily, dosage adjusted based on body weight: 800 mg for < 55 kg, 1200 mg for ≥ 55-75 kg, and 1600 mg for > 75 kg, administered for the first 8 weeks.
  Interventions: Drug: Rifampin; Drug: Isoniazid; Drug: Pyrazinamide; Drug: Ethambutol
- Short-course regimen (Experimental): Drug: Rifapentine, once daily, dosage adjusted based on body weight: 750 mg for ≤41.2 kg, 900 mg for >41.3-48.7 kg, 1050 mg for > 48.8-56.2 kg, 1200 mg for ≥ 56.3 kg, administered for 26 weeks.
  Drug: Moxifloxacin, once daily, 400 mg, administered for 26 weeks. Drug: Isoniazid, once daily, 300 mg, administered for 26 weeks. Drug: Pyrazinamide, once daily, dosage adjusted based on body weight: 1000 mg for < 55 kg, 1500 mg for ≥ 55-75 kg, and 2000 mg for >75 kg, administered for the first 8 weeks.
  Interventions: Drug: Isoniazid; Drug: Rifapentine (RPT); Drug: Moxifloxacin; Drug: Pyrazinamide

INTERVENTIONS:
Drug: Rifampin — Rifampin: once daily, 600 mg.
  Arms: Empirical long course regimen
Drug: Isoniazid — Isoniazid: once daily, 300 mg.
Drug: Rifapentine (RPT) — Rifapentine: once daily with dosage adjusted based on body weight: 750 mg for ≤41.2 kg, 900 mg for >41.3-48.7 kg, 1050 mg for > 48.8-56.2 kg, 1200 mg for ≥ 56.3 kg.
  Arms: Short-course regimen
Drug: Moxifloxacin — Moxifloxacin: once daily, 400 mg.
  Arms: Short-course regimen
Drug: Pyrazinamide — Pyrazinamide: once daily with dosage adjusted based on body weight: 1000 mg for < 55 kg, 1500 mg for ≥ 55-75 kg, and 2000 mg for >75 kg.
Drug: Ethambutol — Ethambutol: once daily with dosage adjusted based on body weight: 800 mg for < 55 kg, 1200 mg for ≥ 55-75 kg, and 1600 mg for > 75 kg.
  Arms: Empirical long course regimen

SUMMARY:
To evaluate the non-inferiority in efficacy between the rifapentine- and moxifloxacin-containing short-course regimens (with rifampicin replaced by rifapentine and ethambutol replaced by moxifloxacin, while isoniazid and pyrazinamide remaining the same as the empirical regimen) and the empirical long-course regimen, so as to determine whether it is possible to shorten the treatment duration to 26 weeks for patients with mild spinal tuberculosis.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 12 years.
2. Based on the medical history, clinical manifestations, radiological, laboratory tests and possible histological samples, the diagnostic criteria are met and judged to be mild spinal tuberculosis.
3. Laboratory test values are completed within 14 days prior to screening.
4. Women of child-bearing potential who are not surgically sterilized must agree to practice a barrier method of contraception or abstain from heterosexual intercourse during study drug treatment.
5. For women of childbearing potential, a negative pregnancy test at or within seven (7) days prior to screening.
6. Karnofsky score greater than or equal to 60.
7. A verifiable address or residence location that is readily accessible for visiting, and willingness to inform the study team of any change of address during the treatment and follow-up period.
8. Written informed consent.

Exclusion Criteria:

- Exclusions Before Randomization:

1. Pregnant or breast-feeding.
2. Unable to take oral medications.
3. Previously enrolled in similar studies.
4. With spinal tumors or metastatic tumors.
5. Patients with mental disorders and cognitive dysfunction.
6. Received any investigational drug in the past 3 months.
7. More than five (5) days of treatment directed against active tuberculosis within 6 months preceding initiation of study drugs.
8. More than five (5) days of systemic treatment with any one or more of the following drugs within 30 days preceding initiation of study drugs: Isoniazid, rifampin, rifambutin, rifabentine, ethambutol, pyrazinamide, kanamycin, amikacin, streptomycin, capreomycin, moxifloxacin, levofloxacin, gatifloxacin, ofloxacin, ciprofloxacin, other fluoroquinolones, ethionamide, prothionamide, cycloserine, terizidone, para-aminosalicylic acid, linezolid, clofazimine, delamanid or bedaquiline.
9. Known history of prolonged QT syndrome.
10. Weight less than 40.0 kg.
11. Known allergy or intolerance to any of the study medications.
12. Individuals will be excluded from enrollment if, at the time of enrollment, their M. tuberculosis isolate is already known to be resistant to any one or more of the following: rifampin, isoniazid, pyrazinamide, ethambutol, or fluoroquinolones.
13. Other medical conditions, that, in the investigator's judgment, make study participation not in the individual's best interest.

    * Exclusions After Randomization:
14. No M. tuberculosis is identified in the screening, baseline, and week 2 samples.
15. Mycobacterium tuberculosis grown from or tested by molecular assays (Xpert MTB / RIF) in samples obtained before or after the study are determined to be resistant to isoniazid, rifampicin, or fluoroquinolones.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-04-05 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
TB-recurrence rate of spinal tuberculosis at 24 months after completion of treatment. | 24 months after completion of treatment
  The recurrence of spinal tuberculosis is defined by the reappearance of pain, with or without sinus formation, loosening or displacement of internal fixation on X-ray, and confirmed by postoperative CT or MRI showing increased local abscess, bone graft absorption, new sequestrum formation, or aggravated bone destruction.
The proportion of participants with grade 3 or more adverse events during study medication | Throughout the study drug treatment period, about 36 months

SECONDARY OUTCOMES:
Clinical cure at the end of therapy | At the end of therapy, WEEK 52 for empirical long-course regimen, WEEK 26 for Short-course regimen
  Clinical Healing: Spinal symptoms improved; pre-disease function restored; weight gain; no instability/neuro deficits.
  Radiological Healing: Reduced epidural/paraspinal abscess/granulation; marrow reconversion; fatty bone reconstitution.
TB-recurrence rate of spinal tuberculosis 12 months after completion of treatment | 12 months after completion of treatment
The proportion of participants who are culture negative at eight weeks | At the end of 8 weeks of treatment
The proportion of discontinuation of assigned treatment for a reason other than microbiological ineligibility | Throughout the study period, an average of 1 year, up until the point of treatment discontinuation due to reasons other than microbiological failure
The incidence of adverse events | Throughout the study drug treatment period, about 36 months
The proportion of participants who have residual neurological dysfunction | Throughout the study drug treatment period, about 36 months
PK parameters of the anti-TB drugs | At the end of therapy, WEEK 52 for empirical long-course regimen, WEEK 26 for Short-course regimen
  Maximum Plasma Concentration [Cmax], etc
PD target attainment rate of the anti-TB drugs | At the end of therapy, WEEK 52 for empirical long-course regimen, WEEK 26 for Short-course regimen
  Cmax/MIC, etc

CONTACTS AND LOCATIONS:
Overall Officials: Wei Zhao, Ph.D, Principal Investigator — Shandong University
Locations (1):
- Shandong Public Health Clinical Center, Jinan, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Wu YE, Cao J, Wang L, Wei YJ, Liu HX, Qi L, Zhang W, Liu F, Zhu ZJ, Fan XT, Wang S, Chen C, Liu XZ, Li Y, Sun ZZ, Pan JB, Yang CQ, Van Den Anker J, Zhang Q, Zhao W. Rifapentine- and moxifloxacin-containing short-course regimens for mild spinal tuberculosis: study protocol for a multicenter, randomized, non-inferiority phase II clinical trial. Front Pharmacol. 2025 Dec 19;16:1684771. doi: 10.3389/fphar.2025.1684771. eCollection 2025. PMID 41487489